CLINICAL TRIAL: NCT05499299
Title: The Effect of Optimised Online Advertising on the Uptake of COVID-19 Vaccines in Hong Kong
Brief Title: Volatility and Heterogeneity of Vaccine Sentiments Means Continuous Monitoring is Needed When Measuring Message Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UW21-428
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Vaccine-Preventable Diseases; Vaccine Refusal
Keywords: Vaccine hesitancy; Google ads; Vaccine messages; Vaccine confidence
MeSH Terms: conditions — Vaccine-Preventable Diseases; Vaccination Refusal; Vaccination Hesitancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Government (Active Comparator): Participants were shown with the government slogan for the COVID-19 vaccine campaign in 2021. This was the control arm.
  Interventions: Behavioral: Google ads
- Comparison (Experimental): The ad emphasized that vaccine uptake in Hong Kong substantially lagged behind that in comparable populations such as Singapore and the UK.
  Interventions: Behavioral: Google ads
- Exemption (Experimental): The ad emphasized that vaccinated people could be exempted from some disruptive control measures such as mandatory testing
  Interventions: Behavioral: Google ads
- Family (Experimental): The ad prompted people to get vaccinated in order to protect their family.
  Interventions: Behavioral: Google ads
- Lottery (Experimental): The ad prompted people to get vaccinated in order to be eligible for the numerous COVID-19 lotteries in Hong Kong
  Interventions: Behavioral: Google ads
- Mortality (Experimental): The ad emphasized that COVID-19 has caused millions of deaths worldwide.
  Interventions: Behavioral: Google ads
- Reopen (Experimental): The ad prompted people to get vaccinated to help Hong Kong reopen sooner.
  Interventions: Behavioral: Google ads

INTERVENTIONS:
Behavioral: Google ads — Individuals who googled COVID-19 information in Hong Kong were randomized to see one of the seven ads and, if they clicked on the ads, the corresponding vaccine message on our website

SUMMARY:
The success of vaccination programs often depends on the effectiveness of the vaccine messages, particularly during emergencies such as the COVID-19 pandemic. The current suboptimal uptake of COVID-19 vaccines across many parts of the world highlights the tremendous challenges in overcoming vaccine hesitancy and refusal even in the context of a world-devastating pandemic. The investigators conducted a randomized controlled trial in Hong Kong to evaluate the impact of seven vaccine messages on COVID-19 vaccine uptake (with the government slogan as the control). The participants included 127,000 individuals who googled COVID-19-related information during July-October 2021.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of using the Google advertising platforms on influencing the uptake of COVID-19 vaccines in Hong Kong. When completed, the rich database compiled through this proposed study will provide increased insight into vaccine hesitancy in Hong Kong. Insights from the optimised online advertising trial can aid in providing crucial technical and theoretical support to the relevant health authorities for any potential evidence-based policy intervention in addressing vaccine hesitancy issues or the public's concerns towards vaccines in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* General users of Google search in Hong Kong

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 127000 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Number of bookings following each message delivery within 6 hours | 6 hours
  The number of bookings made within X = 6 hours following each message delivery

SECONDARY OUTCOMES:
Number of bookings following each message delivery within 3 hours | 3 hours
  The number of bookings made within X = 3 hours following each message delivery
Number of bookings following each message delivery within 12 hours | 12 hours
  The number of bookings made within X = 12 hours following each message delivery

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T Wu, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Proposals should be directed to kathysleung@connect.hku.hk; to gain access, data requestors will need to sign a data access agreement
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal for meta-analysis. Proposals should be directed to Kathyleung@connect.hku.hk; to gain access, data requestors will need to sign a data access agreement.